CLINICAL TRIAL: NCT01925807
Title: Brief Group Intervention for Adolescents With Mild to Moderate Suicidal Ideation and Their Caregivers: Preliminary Investigation for a Novel Treatment Approach
Brief Title: Building Resilience and Attachment in Vulnerable Adolescents
Acronym: BRAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allison Kennedy (Other)
Collaborators: Mach Gaensslen Foundation (Other); AFP Innovation Fund (Other)
Responsible Party: Sponsor-Investigator, Allison Kennedy, Psychologist, Children's Hospital of Eastern Ontario
Organization: Children's Hospital of Eastern Ontario (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHAMO_SI_Group_001
Record Dates: First submitted 2013-08-14; First posted 2013-08-20 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Suicidal Ideation
Keywords: Adolescent; Suicidal Ideation; Emergency Department; Crisis; Attachment; Coping
MeSH Terms: conditions — Suicidal Ideation; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group Intervention (Experimental): The intervention will consist of 6 psycho-educational group sessions for caregivers and 6 psycho-educational group sessions for adolescents. Adolescent and caregiver sessions will be held separately and will focus on different issues. For adolescents, the group sessions will focus on coping strategies and emotional regulation. For caregivers, the group sessions will be focused on attachment, family environment, and validation.
  Interventions: Behavioral: Group Intervention

INTERVENTIONS:
Behavioral: Group Intervention — The intervention will consist of 6 psycho-educational group sessions for caregivers and 6 psycho-educational group sessions for adolescents. Adolescent and caregiver sessions will be held separately and will focus on different issues. For adolescents, the group sessions will focus on coping strategies and emotional regulation. For caregivers, the group sessions will be focused on attachment, family environment, and validation.

SUMMARY:
Suicide is the second leading cause of mortality for Canadian adolescents. Mental health complaints are one of the leading reasons for an emergency department visit at the Children's Hospital of Eastern Ontario and 60% of adolescents report suicidal ideation. The goal of the present investigation is to test the efficacy of a brief group intervention for adolescents with passive suicidal ideation and their caregivers that will focus on coping, familial support, and emotional regulation. The investigators hypothesize that a brief group intervention, delivered in the weeks following presentation for crisis services, will reduce suicidal ideation and improve coping and familial support.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate suicidal ideation
* Recently presented for services in response to a psycho-social crisis (Emergency Department, MH Urgent Care)
* One or two caregiver(s) committed to attending the majority of sessions

Exclusion Criteria:

* Presence of a suicidal plan and/or recent gesture/attempt
* Psychosis
* Schizophrenia
* Dual diagnosis
* Developmental disability or delay
* "Behavioural problem" as primary concern
* Major substance abuse
* Currently receiving mental health services (once every two weeks or more frequently)
* Inability to commit to majority of sessions (minimum 4 of 6 sessions)
* Children's aid society involvement
* Inability of at least one caregiver to commit to attending the majority of sessions

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2014-02; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Suicidal Ideation | 6 weeks
  Suicidal ideation will be measured using the Suicidal Ideation Questionnaire Junior (SIQ-JR; Reynolds, 1988).
  Repeated Measures ANOVA or ANCOVA will be used to compare differences in suicidal ideation within groups (pre-post changes). Further comparisons using clinical cut-off will be conducted via McNemar test for matched pairs.

SECONDARY OUTCOMES:
Familial Support | 6 weeks
  Familial support will be measured using questionnaires for both caregivers and youth. Youth will respond to the Family Environment Scale (Koren, DeChillo, & Friesen, 1992) and the Inventory of Parent and Peer Attachment (Armsden & Greenberg, 1987). Caregivers will respond to the Family Environment Scale and and Relationship Scale Questionnaire (Griffine & Gartholomew, 1994).
  Repeated Measures ANOVA or ANCOVA will be used to compare differences within groups (pre-post changes).

OTHER OUTCOMES:
Coping Strategies | 6 weeks
  Youth coping strategies will be measured using the Youth Stress and Coping Questionnaire (Cloutier et al., 2008).
  Repeated Measures ANOVA or ANCOVA will be used to compare differences within groups (pre-post changes).
Depression | 6 weeks
  Youth depression will be measured using the Children's Depression Inventory-2 Self report (CDI-2; Kovaks, 2010).
  Repeated Measures ANOVA or ANCOVA will be used to compare differences within groups (pre-post changes).
Anxiety | 6 weeks
  Youth anxiety symptoms will be measured using the Multidimensional Anxiety Scale for Children (MASC-2; March, 1997).
  Repeated Measures ANOVA or ANCOVA will be used to compare differences within groups (pre-post changes).

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kennedy, Ph.D., Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Diamond GS, Wintersteen MB, Brown GK, Diamond GM, Gallop R, Shelef K, Levy S. Attachment-based family therapy for adolescents with suicidal ideation: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2010 Feb;49(2):122-31. doi: 10.1097/00004583-201002000-00006. PMID 20215934
- [Background] Rathus JH, Miller AL. Dialectical behavior therapy adapted for suicidal adolescents. Suicide Life Threat Behav. 2002 Summer;32(2):146-57. doi: 10.1521/suli.32.2.146.24399. PMID 12079031
- [Background] Armsden GC, Greenberg MT. The inventory of parent and peer attachment: Individual differences and their relationship to psychological well-being in adolescence. J Youth Adolesc. 1987 Oct;16(5):427-54. doi: 10.1007/BF02202939. PMID 24277469
- [Background] Cloutier, P. F., Kennedy, A., & Glennie, E. (2008, June). Coping behaviors and intensity of non-suicidal self-harm in Canadian adolescents presenting to emergency mental health services. Poster presented at the third annual meeting of the International Society for the Study of Self-Injury (ISSS), Harvard University, Cambridge, MA.
- [Background] Kovacs, M. (2010). Children's Depression Inventory Manual. Toronto, ON: Multi-Health Systems Inc.
- [Background] March, J.S. (2013). Manual for the Multidimensional Anxiety Scale for Children - 2nd Edition (MASC-2). Toronto, ON: MHS Inc.
- [Background] Moos, R. H., & Moos, B. S. (1981). Family environment scale manual
- [Background] Reynolds, W. M. (1988). Suicidal Ideation Questionnaire Professional Manual (p. 47).
- [Background] Griffine, D. W., & Garthholomew, K. (1994). The metaphysics of measurement: The case of adult attachment. (pp. 17-52).